CLINICAL TRIAL: NCT06669546
Title: Preventing Cognitive Decline Using Portable, Non-invasive Sleep Enhancement
Brief Title: Effects of Real vs. Soundless Acoustic Stimulation During Deep Sleep on Brain Activity, Memory, and Blood Biomarkers in Older Adults (60-85) With Mild Memory Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Zurich (Other); Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-00409; 215333 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Decline; Alzheimer Disease; Subjective Cognitive Decline (SCD); Mild Cognitive Impairment (MCI); Cognitive Impairment, Mild
Keywords: Sleep; Dementia; Prevention; Phase-locked auditory stimulation; Blood-based biomarkers; Home; Longitudinal; Electroneurophysiology; EEG; Memory; Cognition; Serious games; Old age; Human
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia | interventions — Acoustic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLAS first, sham second (Experimental): In this study arm, participants will undergo a 4-week intervention period with real phase-locked auditory stimulation (PLAS) administered on nights from Monday to Friday. Following this initial intervention period, participants will have a 2-week washout phase. Finally, participants will enter the second intervention period, during which sham (soundless) PLAS will be administered.
  Interventions: Other: Phase-locked auditory stimulation (PLAS); Other: Sham Phase-Locked Auditory Stimulation
- Sham first, PLAS second (Experimental): In this study arm, participants will undergo a 4-week intervention period with sham (soundless) phase-locked auditory stimulation (PLAS) administered on nights from Monday to Friday. Following this initial intervention period, participants will have a 2-week washout phase. Finally, participants will enter the second intervention period, during which real PLAS will be administered.
  Interventions: Other: Phase-locked auditory stimulation (PLAS); Other: Sham Phase-Locked Auditory Stimulation

INTERVENTIONS:
Other: Phase-locked auditory stimulation (PLAS) — Intervention: Verum Phase-Locked Auditory Stimulation (PLAS) Using the SleepLoop Device.
  The experimental intervention utilizes the SleepLoop device, a home-use, EEG-based system designed for phase-locked acoustic stimulation (PLAS). The device continuously monitors sleep through EEG (Fpz) alongside electrooculogram (EOG) and electromyogram (EMG) channels. The device employs a closed-loop algorithm that detects slow oscillations (SOs) in the EEG and delivers short sound stimuli (50 ms pink noise) during the positive half-waves of slow waves in slow-wave sleep (SWS). These stimuli are delivered through integrated headphones in the SleepLoop device. The intervention is applied during work days for 4 weeks. The algorithm is only active during SWS and does not deliver stimuli when the participant is awake, or in lighter sleep stages (N1, N2) or REM sleep. The intensity and algorithm sensitivity are individually calibrated for each participant to optimize stimulation.
  Other Names: Acoustic stimulation; Phase-targeted auditory stimulation (PTAS); Auditory stimulation; Closed-loop acoustic stimulation
Other: Sham Phase-Locked Auditory Stimulation — Participants will undergo the same procedure as the real Phase-Locked Auditory Stimulation (PLAS) intervention. However, during the sham condition, the headphones are turned off, and no auditory stimulation is delivered.

SUMMARY:
This study aims to explore a non-invasive way to improve memory and slow cognitive decline in older adults by enhancing sleep quality. Dementia, a leading cause of death worldwide, is often associated with disturbed sleep, particularly the loss of deep, slow-wave sleep (SWS). SWS is important for memory and clearing waste from the brain. Poor SWS can worsen memory loss and allow harmful waste to build up, which may increase the risk of dementia.

The investigators are testing whether phase-locked auditory stimulation (PLAS) can improve SWS in people at a mild stage of cognitive impairment. PLAS uses short sounds played at specific moments to strengthen slow-wave brain activity during sleep. The investigators previous laboratory based research has shown that this can improve memory and help with clearing waste from the brain. Now, the investigators want to test this in a real-world setting, over a longer period, which is unfeasible in a laboratory setting.

In this study, 60 older adults will use home-use devices that deliver either real or sham (soundless) PLAS across two different 4-week periods. Memory will be tested using engaging "serious games." Before and after each experimental period, blood samples will be taken to measure dementia-related markers, and cognitive batteries will be performed. The investigators expect that PLAS will improve sleep, and that this will have a downstream effect on memory and brain clearance, potentially slowing the process of cognitive decline.

If successful, this could lead to the development of an affordable treatment that helps people maintain brain health and prevent dementia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age between 60 and 85 years
* Cognitive impairment (subjective and/or MoCA between 23-26)
* Native German speakers or comparably fluent
* Normal or corrected-to-normal vision.
* Intact hearing
* A close cohabitant (partner/sibling) should be present to support participants in using study materials/devices.

Exclusion Criteria:

* Insomnia assessed by the Regensburg Insomnia Scale (RIS; Crönlein et al., 2013)
* Restless leg syndrome assessed by questions concerning typical symptoms.
* Sleep apnoea assessed by the Berlin Questionnaire (BQ; Netzer et al., 1999)
* Severely irregular sleep patterns assessed by the RIS and the Pittsburgh sleep quality index (PSQI; Buysse et al., 1989)
* Symptoms of depression (Geriatric Depression Scale (GDS; Yesavage et al., 1982) ≥ 5)
* History of untreated severe neurological and psychiatric diseases
* Alcohol or substance abuse
* Use of medication acting on the central nervous system

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Episodic memory performance differences (between and within subject) according to the experimental condition | Participants will play serious games on weekdays during the adaptation week, as well as on weekdays throughout both the first and second 4-week intervention periods.
  Episodic memory performance will be assessed by means of serious games.

SECONDARY OUTCOMES:
Electrophysiological Response - Event-Related Potentials (ERPs) | Sleep-Electrophysiology will be measured on weekdays during the adaptation week, as well as on weekdays throughout both the first and second 4-week intervention periods.
  Electrophysiological responses will be measured via EEG to assess event-related potentials (ERPs) in response to real versus sham acoustic stimulation.
Electrophysiological Response - Power, Number, and Amplitude of Slow Oscillations (SO) and Spindles | Sleep-electrophysiology will be measured on weekdays during the adaptation week, as well as on weekdays throughout both the first and second 4-week intervention periods.
  Electrophysiological responses will be measured via EEG to assess the power, number, and amplitude of slow oscillations (SO) and sleep spindles in response to real versus sham acoustic stimulation.
Electrophysiological Response - Coupling of Slow Oscillations and Sleep Spindles | Sleep-electrophysiology will be measured on weekdays during the adaptation week, as well as on weekdays throughout both the first and second 4-week intervention periods.
  Electrophysiological responses will be measured via EEG to assess the coupling between slow oscillations and spindles in response to real versus sham acoustic stimulation.
Amyloid-Beta Response | At baseline, after 4 weeks, after 6 weeks, after 10 weeks
  Blood samples will be collected to measure plasma amyloid-beta levels and compare them across conditions.
Electrophysiology - Brain Age Estimation | Sleep electrophysiology will be measured on weekdays during the adaptation week and on weekdays throughout both the first and second 4-week intervention periods.
  EEG, EMG, and ECG will be used to estimate brain age and assess whether PLAS leads to a rejuvenation of the brain, reflecting a younger brain state. Machine learning will analyze sleep-EEG data to provide an accurate brain age estimate.

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Züst, PhD, Principal Investigator — University Hospital of Old Age Psychiatry and Psychotherapy, University of Bern, 3000 Bern, Switzerland
Locations (1):
- University Hospital of Old Age Psychiatry and Psychotherapy, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Currently, there are no collaborations to disclose, but the investigators are generally open to such endeavours in the future. For this purpose, general consent for reuse of data is being collected from participants.

REFERENCES:
- [Background] Lustenberger C, Ferster ML, Huwiler S, Brogli L, Werth E, Huber R, Karlen W. Auditory deep sleep stimulation in older adults at home: a randomized crossover trial. Commun Med (Lond). 2022 Apr 4;2:30. doi: 10.1038/s43856-022-00096-6. eCollection 2022. PMID 35603302
- [Background] Wunderlin M, Zust MA, Hertenstein E, Feher KD, Schneider CL, Kloppel S, Nissen C. Modulating overnight memory consolidation by acoustic stimulation during slow-wave sleep: a systematic review and meta-analysis. Sleep. 2021 Jul 9;44(7):zsaa296. doi: 10.1093/sleep/zsaa296. PMID 33406249
- [Background] Zeller CJ, Wunderlin M, Wicki K, Teunissen CE, Nissen C, Zust MA, Kloppel S. Multi-night acoustic stimulation is associated with better sleep, amyloid dynamics, and memory in older adults with cognitive impairment. Geroscience. 2024 Dec;46(6):6157-6172. doi: 10.1007/s11357-024-01195-z. Epub 2024 May 14. PMID 38744792
- [Background] Wunderlin M, Zeller CJ, Senti SR, Feher KD, Suppiger D, Wyss P, Koenig T, Teunissen CE, Nissen C, Kloppel S, Zust MA. Acoustic stimulation during sleep predicts long-lasting increases in memory performance and beneficial amyloid response in older adults. Age Ageing. 2023 Dec 1;52(12):afad228. doi: 10.1093/ageing/afad228. PMID 38163288
- See also: Information on current sleep studies at the Memory Clinic Bern, focused on research related to sleep and cognitive function. — https://www.memory-clinic-bern.ch/aktuelle-studien/schlafstudie/